CLINICAL TRIAL: NCT03524066
Title: Understanding the Lung Pharmacokinetics (PK) in Humans by Direct Sampling of Epithelial Lining Fluid (ELF) After Inhalation and Oral Administration of Model Drugs
Brief Title: Lung Pharmacokinetics (PK) in Epithelial Lining Fluid (ELF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17-15 BROSO
Record Dates: First submitted 2018-04-25; First posted 2018-05-14 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Healthy
MeSH Terms: interventions — Inhalation; Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhaled + Bronchoscopy (Experimental): One-time Inhalation of Salbutamol 200 µg, Salmeterol 50µg and Fluticasone 500µg. During two bronchoscopic procedures two pre-specified lung tissue sites (middle lobe and lingula) will be sampled. Bronchoadsorption sample, bronchial brushing, mucosal biopsy, and bronchoalveolar lavage (BAL) samples will be taken from each site.
  Interventions: Drug: Inhalation; Other: Bronchoscopy
- Systemic + Bronchoscopy (Experimental): One-time Salbutamol (8 mg) and Propranolol (40mg) administered orally. During two bronchoscopic procedures two pre-specified lung tissue sites (middle lobe and lingula) will be sampled. Bronchoadsorption sample, bronchial brushing, mucosal biopsy, and BAL samples will be taken from each site.
  Interventions: Drug: Systemic; Other: Bronchoscopy

INTERVENTIONS:
Drug: Inhalation — Salbutamol(200µg), Salmeterol (50µg) and Fluticasone propionate (500µg) by inhalation
  Arms: Inhaled + Bronchoscopy
Drug: Systemic — Salbutamol 8mg M/R Tablet, Propranolol 40 mg administered orally
  Arms: Systemic + Bronchoscopy
Other: Bronchoscopy — Bronchoadsorption sample, bronchial brushing, mucosal biopsy, and BAL samples during bronchoscopy

SUMMARY:
The aim of the present study is to increase the general understanding of lung PK of selected compounds by sampling epithelial lining fluid ELF and lung tissue.

DETAILED DESCRIPTION:
This study will investigate drug levels of selected compounds at multiple sites in the lung and explore different innovative sampling methods to obtain information on lung PK. The aim of the study is not to generate safety or efficacy data of the selected licensed drugs. The choice of drugs is based on general considerations regarding therapy of airway diseases and the physical-chemical properties of the compounds. It is not driven by the compounds per se.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, aged 18-50 years. Women will be considered for inclusion if they are: Not pregnant, as confirmed by pregnancy test (see flow chart), and not nursing. Of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal, with documented proof of hysterectomy or tubal ligation, or meets clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the screening visit). Of childbearing potential and using a highly effective method of contraception during the entire study (vasectomised partner, sexual abstinence - the lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to the first dose of study medication until at least 72 hours after treatment -, implants, injectables, combined oral contraceptives, hormonal IUDs (Intrauterine devices) or double-barrier methods, i.e. any double combination of IUD, condom with spermicidal gel, diaphragm, sponge, and cervical cap).
* Normal lung function with Forced Expiratory Volume in the first second (FEV1) predicted ≥ 80% and FEV1/Forced Vital Capacity (FVC) > 70%.
* Nonsmokers with a history of less than 1 pack year having been nonsmokers for at least the last five years
* Body mass index between 18 and 32 kg/m²
* Able and willing to give written informed consent.

Exclusion Criteria:

* Past or present disease, which as judged by the investigator, may affect the outcome of the study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, psychiatric disease, endocrine disease, infectious disease, inflammatory disease or pulmonary disease (including but not confined to asthma, tuberculosis, bronchiectasis or cystic fibrosis)
* Regular intake of any prescribed or over the counter medication. Exceptions include paracetamol for pain relief, oral contraceptive medication, hormonal replacement therapy, dietary and vitamin supplements
* Clinically relevant history of allergy as judged by the investigator
* Intolerance or contraindications to medications applied as model drugs (e.g. hyperthyreosis) or for sedation during bronchoscopy
* Infections of the lower respiratory tract within 4 weeks before visit 1, visit 2, or visit 3. These patients can be rescreened starting from visit 1.
* Any clinically relevant abnormal findings in physical examination, clinical chemistry, hematology, urinalysis, vital signs, lung function, or ECG at Visit 1, which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or may influence the results of the study, or the subject's ability to participate in the study
* History of drug or alcohol abuse
* Risk of non-compliance with study procedures
* Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Maximum concentration of Salbutamol in the lung | change from baseline to 1 hour and 24,5 hours post dose
  Maximum concentration of Salbutamol in samples from bronchoscopy (bronchoadsorption, bronchial brushing, mucosal biopsy, Bronchoalveolar lavage (BAL))
Maximum concentration of Salmeterol in the lung | change from baseline to 1 hour and 24,5 hours post dose
  Maximum concentration of Salmeterol in samples from bronchoscopy (bronchoadsorption, bronchial brushing, mucosal biopsy, Bronchoalveolar lavage (BAL))
Maximum concentration of Fluticasone in the lung | change from baseline to 1 hour and 24,5 hours post dose
  Maximum concentration of Fluticasone in samples from bronchoscopy (bronchoadsorption, bronchial brushing, mucosal biopsy, Bronchoalveolar lavage (BAL))
Maximum concentration of Propranolol in the lung | change from baseline to 1 hour and 24,5 hours post dose
  Maximum concentration of Propranolol in samples from bronchoscopy (bronchoadsorption, bronchial brushing, mucosal biopsy, Bronchoalveolar lavage (BAL))

SECONDARY OUTCOMES:
Maximum concentration of Salbutamol in plasma | change from baseline to 0,25 hour (h) 0,5 h, 1 h, 2 h, 4h, 8 h, 12 h, 24 h, 36 h, 48 h post dose
  Maximum concentration of Salbutamol in plasma samples
Maximum concentration of Salmeterol in plasma | change from baseline to 0,25 hour (h) 0,5 h, 1 h, 2 h, 4h, 8 h, 12 h, 24 h, 36 h, 48 h post dose
  Maximum concentration of Salmeterol in plasma samples
Maximum concentration of Fluticasone in plasma | change from baseline to 0,25 hour (h) 0,5 h, 1 h, 2 h, 4h, 8 h, 12 h, 24 h, 36 h, 48 h post dose
  Maximum concentration of Fluticasone in plasma samples
Maximum concentration of Propranolol in plasma | change from baseline to 0,25 hour (h) 0,5 h, 1 h, 2 h, 4h, 8 h, 12 h, 24 h, 36 h, 48 h post dose
  Maximum concentration of Propranolol in plasma samples

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hohlfeld, MD, Principal Investigator — Fraunhofer ITEM
Locations (1):
- Fraunhofer Institute for Toxicology and Experimental Medicine, Hanover, Germany